CLINICAL TRIAL: NCT01700673
Title: A Phase II Study of 5-Azacitidine (5AC) in Combination With Sargramostim (GM-CSF) as Maintenance Treatment, After Definitive Therapy With Either Stem Cell Transplant (SCT) or Cytarabine-based Chemotherapy, in Patients With Poor-risk Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: Phase II Study of Azacitidine and Sargramostim as Maintenance Treatment for Poor-Risk AML or MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1240; P01CA015396 (NIH); NA_00072223 (Other: JHMIRB)
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2021-08

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: maintenance treatment; stem cell transplant; cytarabine-based chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Myeloablative BMT (Experimental): Azacitidine and sargramostim after myeloablative stem cell transplant
  Interventions: Drug: Azacitidine; Biological: Sargramostim
- Non-myeloablative BMT (Experimental): Azacitidine and sargramostim after non-myeloablative stem cell transplant
  Interventions: Drug: Azacitidine; Biological: Sargramostim
- Standard consolidation (Experimental): Azacitidine and sargramostim after standard consolidation
  Interventions: Drug: Azacitidine; Biological: Sargramostim

INTERVENTIONS:
Drug: Azacitidine — Azacitidine will be administered days 1-5 of a 28 day cycle. Treatment is planned for a total of 12 cycles.
  Other Names: Vidaza; 5-azacytidine; Azacytidine
Biological: Sargramostim — Sargramostim will be administered days 1-10 of a 28 day cycle. Treatment is planned for a total of 12 cycles.
  Other Names: GM-CSF

SUMMARY:
To determine the impact of maintenance therapy in patients with MDS/AML in remission.

DETAILED DESCRIPTION:
We propose a phase II study to determine the impact of maintenance therapy with 5-azacytidine and GM-CSF in patients with poor-risk AML or MDS, who are in remission after definitive treatment with either stem cell transplant or cytarabine-based consolidation chemotherapy.

In order to precede relapse and to avoid lead time bias, treatment would need to commence within 185 days of definitive therapy. Furthermore, approximately 50% of relapses occur within the first year and up to 80% within two years after SCT, therefore we would limit the duration of maintenance therapy to one year, followed by two years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 6 months
2. Initial diagnosis of poor -risk AML or MDS (defined in section 3.2), treated with either stem cell transplant or cytarabine-based consolidation chemotherapy, within the past 60-185 days
3. ECOG performance status 0-2
4. No morphologic evidence of leukemia or active MDS as determined by JHH Hematopathologist independent review of a bone marrow aspirate and biopsy done following the completion of therapy and within 14 days prior to enrollment
5. Peripheral blood count recovery: Neutrophil count ≥ 1000 /µL, platelet count ≥ 50x 109 /µL without platelet transfusions, and adequate hematocrit independent of red cell transfusions .
6. No evidence of extramedullary leukemia, such as CNS or soft tissue involvement
7. Adequate end organ function as measured by the following: AST and ALT < 4 x normal, total serum bilirubin < 2 x upper limit normal (unless due to hemolysis, Gilbert's syndrome, or ineffective erythropoiesis), creatinine < 2 x upper limit of normal
8. Ability to give informed consent
9. In agreement to use an effective barrier method of birth control to avoid pregnancy during the study and for a minimum of 30 days after study treatment, for all male and female patients who are fertile

Exclusion Criteria:

1. Patients with untreated or uncontrolled infections
2. Patients with untreated or uncontrolled grade 3 or 4 GVHD
3. Pregnancy and lactation
4. Concurrent use of any other investigational agents.
5. Known HIV-positive patients.
6. Known hypersensitivity to 5AC or GM-CSF

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Showel, MD, Study Chair — JHU
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Myeloablative BMT | Non-myeloablative BMT | Standard Consolidation
Started | 1 | 23 | 1
Completed | 1 | 17 | 1
Not Completed | 0 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Myeloablative BMT | Non-myeloablative BMT | Standard Consolidation | Total
Number analyzed (Participants) | 1 | 23 | 1 | 25
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 72 years | 1 | 23 | 1 | 25
  >=73 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 11 | 1 | 12
  Male | 1 | 12 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 1 | 18 | 1 | 20
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Two-year Relapse Free Survival of Patients
Description: To evaluate the two-year relapse-free survival (RFS) of patients with poor-risk Acute Myeloid Leukemia (AML) or Myelodysplasia (MDS), who receive maintenance treatment with 5-Azacytidine (5AC) in combination with sargramostim (GM-CSF) during remission, following definitive therapy with either a stem cell transplant (SCT) or cytarabine-based consolidation chemotherapy.
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Non-myeloablative BMT | Myeloablative BMT | Standard Consolidation
Number analyzed (Participants) | 17 | 1 | 1
Participants | 8 | 1 | 1

2. Secondary Outcome: Hematologic Toxicity as Determined by Anemia
Description: Percentage of patients with anemia, the most commonly reported hematologic toxicity, after receiving the combination of Azacitidine and sargramostim
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Non-myeloablative BMT | Myeloablative BMT | Standard Consolidation
Number analyzed (Participants) | 17 | 1 | 1
Participants | 8 | 1 | 0

3. Secondary Outcome: One-year RFS
Description: We will report the number of participants with one year RFS
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Non-myeloablative BMT | Myeloablative BMT | Standard Consolidation
Number analyzed (Participants) | 17 | 1 | 1
Participants | 12 | 1 | 1

4. Secondary Outcome: Overall Survival
Description: Percentage of participants with overall survival at 2 years.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Non-myeloablative: Azacitidine and sargramostim after non-myeloablative stem cell transplant
Arm/Group | Non-myeloablative | Myeloablative BMT | Standard Consolidation
Number analyzed (Participants) | 11 | 1 | 1
Participants | 6 | 1 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Non-myeloablative BMT | Myeloablative BMT | Standard Consolidation
All-Cause Mortality (participants affected / at risk) | 8/17 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 4/17 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 17/17 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-myeloablative BMT (N=17) | Myeloablative BMT (N=1) | Standard Consolidation (N=1)
anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Graft-vs-host disease (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
infections (Infections and infestations) | 4 | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-myeloablative BMT (N=17) | Myeloablative BMT (N=1) | Standard Consolidation (N=1)
nausea (Gastrointestinal disorders) | 8 (13) | 1 | 1 (2)
ALT increase (Blood and lymphatic system disorders) | 3 (12) | 0 | 1
anemia (Blood and lymphatic system disorders) | 8 (21) | 1 | 0
anorexia (Gastrointestinal disorders) | 3 (6) | 0 | 0
edema (Blood and lymphatic system disorders) | 2 (5) | 0 | 1 (2)
myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 | 0
bone pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 0 | 1
chills (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 | 0
constipation (Gastrointestinal disorders) | 4 (16) | 0 | 1
creatinine increase (Blood and lymphatic system disorders) | 2 (5) | 0 | 0
diarrhea (Gastrointestinal disorders) | 8 (15) | 0 | 1
dizziness (Ear and labyrinth disorders) | 4 (6) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 0 | 1
dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (12) | 0 | 0
eosiniphilia (Blood and lymphatic system disorders) | 2 (3) | 0 | 0
injection site erythema (Skin and subcutaneous tissue disorders) | 12 (17) | 1 | 0
fatigue (General disorders) | 9 (27) | 0 | 1
graft-vs-host disease (Skin and subcutaneous tissue disorders) | 4 (9) | 1 | 0
headache (Nervous system disorders) | 6 (8) | 0 | 1
infections (Infections and infestations) | 14 (44) | 0 | 1
insomnia (Nervous system disorders) | 4 (9) | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 8 (19) | 0 | 1 (3)
pruritis (Skin and subcutaneous tissue disorders) | 6 (13) | 0 | 1 (4)
neutropenia (Blood and lymphatic system disorders) | 5 (13) | 0 | 1
leukopenia (Blood and lymphatic system disorders) | 4 (12) | 0 | 1
thrombocytopenia (Blood and lymphatic system disorders) | 8 (23) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT01700673/Prot_SAP_000.pdf